CLINICAL TRIAL: NCT02452177
Title: Preventive and Reversional Effect of Vitamin D on Parenteral Nutrition Associated Liver Disease: Clinical Observation and Experimental Study
Brief Title: Preventive and Reversional Effect of Vitamin D on Parenteral Nutrition Associated Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengxian Fan (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Shengxian Fan, M.D., Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Jinling Hospital
Record Dates: First submitted 2015-05-16; First posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Liver Disease
Keywords: parenteral nutrition associated liver disease; vitamin D; short bowel syndrome; farnesoid X receptor; cholestasis
MeSH Terms: conditions — Liver Diseases; Short Bowel Syndrome; Cholestasis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Experimental): Patients in this group were treated with oral vitamin D at a dose of 1200 IU per day for 2 months.
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator)

INTERVENTIONS:
Drug: Vitamin D
  Arms: Vitamin D

SUMMARY:
Patients who accept long-term parenteral nutrition tend to suffer from liver injury. The mechanism for this injury has two possible explanations. The first possible reason is intrinsic toxic effects of parenteral nutrition. The second is the basic pathological condition of intestinal failure which includes infection, bacterial translocation, etc. Cholestasis is the lethal presentation of this kind of liver disease. Farnesoid X receptor (FXR) is a member of ligand-activated nuclear receptor superfamily. FXR serves as a sensor for bile acids and promotes enterohepatic clearance of bile acids by controlling the expression of genes involved in their transport and metabolism. Considering the activation of vitamin D receptor (VDR) by vitamin D can induce FXR-related genes in the liver.The hypothesis of this study is that vitamin D plays a key role in the prevention and reversion of the liver via VDR and/or FXR signaling pathway. Using a mouse cholestasis model based on short bowel syndrome and parenteral nutrition, the researchers will investigate the dynamic change of plasma vitamin D level. Afterward, intravenous supplement of vitamin D was added to this model to demonstrate vitamin D can ameliorate cholestasis. An in vitro system was developed to investigate the importance of FXR signaling pathway in this effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients with short bowel syndrome supported by total parenteral nutrition.
* Patients have intestine more than 50cm.
* Requirements of informed consent and assent of participant, parent or legal guardian as applicable consciousness and ability cooperate.

Exclusion Criteria:

* Patients have obstruction of biliary tract, infection, autoimmune disease, cancer.
* Patients have intestine less than 50cm.
* A clinically significant laboratory abnormality or a history of significant cardiac, pulmonary, hepatic, or renal disease.
* Female with positive pregnancy.
* Allergy to ursodeoxycholic acid.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-10 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
liver function | two months
  Serum aspartate aminotransferase, alanine aminotransferase (ALT), gamma glutamyl transferase (GGT), triglyceride, very low density lipoprotein (VLDL), and bilirubin (total, direct, and indirect) were analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China